CLINICAL TRIAL: NCT07389408
Title: A Prospective, Multicenter Registry to Observe the Treatment Patterns, Clinical Outcomes, and Decision-Making in Patients With Early Breast Cancer Eligible for EndoPredict® Testing
Acronym: PRELUDE
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Michalis Kontos, Professor in Breast and General Surgery, National and Kapodistrian University of Athens
Other Study IDs: 84/18.03.2025
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Adenocarcinoma
Keywords: breast cancer; luminal subtype; EndoPredict; genetic signature; survival
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-metastatic breast cancer N0-N1 patients eligible for EndoPredict testing: Subjects diagnosed with non-metastatic invasive breast cancer, pT1-pT3, with 0 to 3 positive axillary lymph nodes, ER-positive, HER2-negative, that have not received neo-adjuvant chemotherapy and therefore are eligible for EndoPredict® testing. No intervention is planned, as this is an observational study and treatment of patients will not be changed due to their participation in the study.

SUMMARY:
The study is planned to observe and document the therapeutic decision-making process, treatment protocols, and clinical outcomes in patients with luminal breast cancer, whether they have undergone EndoPredict® testing or not

DETAILED DESCRIPTION:
PRELUDE is a prospective, multicenter, non-interventional registry designed to describe real-world treatment decision-making, treatment patterns, and long-term clinical outcomes in patients with luminal (ER-positive/HER2-negative) early breast cancer who are eligible for EndoPredict® testing, including patients who do and do not undergo the test.

The registry will be conducted at approximately 10-20 sites across Greece (with the option to add sites outside Greece if needed) and aims to enroll up to 2,000 eligible participants within 3 years. Participants may be enrolled after surgical histopathology results are available and before commencement of adjuvant endocrine treatment, and will be followed prospectively once per year for up to 10 years after surgery.

The study aims to assess 5- and 10-year clinical outcomes and to evaluate these outcomes according to EndoPredict® (EP/EPclin) risk groups or scores among patients who undergo testing, in a real-world setting. The registry will also examine which patient and disease characteristics (e.g., age, menopausal status, nodal status, histopathology, EPclin score) will influence adjuvant treatment decisions, in the context of evolving therapeutic standards and recently introduced adjuvant options.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Histological diagnosis of invasive breast cancer.
* T1-T3 tumor size.
* 0-3 positive axillary lymph nodes.
* Documented ER-positive tumor by immunohistochemistry (≥1% or Allred Score: ≥3/8 or H-score: ≥50/ 300)
* Documented HER2-negative tumor by immunohistochemistry and/or in situ hybridization
* Subject with signed and dated informed consent form.

Exclusion Criteria:

* History of another primary malignancy within the last 5 years, except for resected non-melanoma skin cancer.
* Pre-operative chemotherapy administered.
* Subject without signed and dated informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects diagnosed with invasive breast cancer, pT1-pT3, with 0 to 3 positive axillary lymph nodes, ER-positive, HER2-negative, that have not received neo-adjuvant chemotherapy and therefore are eligible for EndoPredict® testing.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Distant relapse free survival (DRFS) | 5- and 10-years
  To collect and evaluate distant relapse-free survival (DRFS) at 5 and 10 years in patients with luminal breast cancer, with analyses stratified by EPclin risk group among participants who undergo EndoPredict® testing.
Overall Survival (OS) | 5- and 10-years
  To collect and evaluate overall survival (OS) at 5 and 10 years in patients with luminal breast cancer, with analyses stratified by EPclin risk group among participants who undergo EndoPredict® testing.
Distant relapse free interval (DRFI) | 5- and 10-years
  To collect and evaluate distant relapse free interval (DRFI) at 5 and 10 years in patients with luminal breast cancer, with analyses stratified by EPclin risk group among participants who undergo EndoPredict® testing.
Proportion of adjuvant chemotherapy administration and association with baseline clinicopathologic characteristics and EPclin score | Up to 2 months post-operatively
  Proportion of participants who received adjuvant chemotherapy (yes/no) and its association with baseline clinicopathologic characteristics (age, menopausal status, nodal status, T stage, N stage, histologic grade) and EPclin score.

SECONDARY OUTCOMES:
Local relapse free survival (LRFS) | 5- and 10-years
  To collect and evaluate local relapse free survival (LRFS) at 5 and 10 years in patients with luminal breast cancer, with analyses stratified by EPclin risk group among participants who undergo EndoPredict® testing.
Performance of EndoPredict (assessed with DRFS) in specific population subgroups [multifocal-multicentric disease (MFMC), node-positive, pre-menopausal women] | 5- and 10-years
  Performance of EndoPredict in specific population subgroups [multifocal-multicentric disease (MFMC), node-positive patients, pre-menopausal women], assessed with distant recurrence free survival (DRFS).
Performance of EndoPredict (assessed with DRFI) in specific population subgroups [multifocal-multicentric disease (MFMC), node-positive, pre-menopausal women] | 5- and 10-years
  Performance of EndoPredict in specific population subgroups [multifocal-multicentric disease (MFMC), node-positive patients, pre-menopausal women], assessed with distant recurrence free interval (DRFI).
OS in specific sub-groups (MFMC, node-positive, pre-menopausal women) | 5- and 10-years
  OS in specific sub-groups (MFMC, node-positive, pre-menopausal women)
DRFS in specific sub-groups (MFMC, node-positive, pre-menopausal women) | 5- and 10-years
  DRFS in specific sub-groups (MFMC, node-positive, pre-menopausal women)
DRFI in specific sub-groups (MFMC, node-positive, pre-menopausal women) | 5- and 10-years
  DRFI in specific sub-groups (MFMC, node-positive, pre-menopausal women)
LRFS in specific sub-groups (MFMC, node-positive, pre-menopausal women) | 5- and 10-years
  LRFS in specific sub-groups (MFMC, node-positive, pre-menopausal women)

CONTACTS AND LOCATIONS:
Locations (13):
- Greece (13):
  - "Elena Venizelou" General Hospital, Department of Surgery, Athens
  - "Prolipsis" Center, Breast Unit, Athens
  - Henry Dunant Hospital Center, 3rd Breast Surgical Department, Athens
  - Laiko Hospital, National and Kapodistrian University of Athens, Medical School, Athens
  - Mediterraneo Hospital, Breast Clinic, Athens
  - Metropolitan General Hospital, 3rd Breast Clinic, Cholargós
  - Metropolitan General Hospital, 4th Breast Clinic, Cholargós
  - "Apollonio-Theotokos" General Clinic, Department of Surgery, Larissa
  - IASO Thessalias General Clinic, Breast Surgery Department, Larissa
  - IASO General Clinic, 2nd Breast Clinic, Marousi
  - MITERA, 1st Breast Clinic, Marousi
  - Thessaloniki Bioclinic Hospital, Breast Unit, Thessaloniki
  - General Hospital of Trikala, Breast Surfery Dept., Trikala

IPD SHARING:
Plan to Share IPD: Undecided